CLINICAL TRIAL: NCT02180230
Title: Immediate Function of NobelSpeedy Shorty and Brånemark System® Mk III Shorty Implants in Daily Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nobel Biocare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T-127
Record Dates: First submitted 2014-06-26; First posted 2014-07-02 (Estimated); Results first posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2015-12

CONDITIONS: Partial Edentulism; Complete Edentulism
Keywords: Short implants; prospective multicenter study; maxilla & mandible

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Shorty implants (Other): Brånemark System Mk III Shorty and/or NobelSpeedy Shorty
  Interventions: Device: Shorty implants

INTERVENTIONS:
Device: Shorty implants — Dental implant insertion to maxilla or mandible
  Other Names: Brånemark System Mk III Shorty and/or NobelSpeedy Shorty

SUMMARY:
The aim of this study was to evaluate the 7 mm long implants NobelSpeedy Shorty and Brånemark System Mk III Shorty: by determining the marginal bone remodeling, implant survival rate, soft tissue health and maintenance.

DETAILED DESCRIPTION:
The primary endpoint was the change in marginal bone levels (in mm) from the time of implant insertion to follow-up visits (3, 6, 12, 36 and 60 months).

Further endpoints were:

* cumulative survival rates of the implants
* soft tissue parameters (papilla index, bleeding on probing)
* plaque formation

ELIGIBILITY:
Inclusion Criteria:

* The subjects should have an osseous architecture enough to receive an implant with a diameter of at least 3.75 mm for Brånemark System Mk III Shorty or 4 mm for NobelSpeedy Shorty and a sufficient amount of bone for placing implants with a length of 7 mm.
* The final tightening torque at installation should be 35-45 Ncm without further rotation and should not exceed 45 Ncm.
* The subject as well as the implant site(s) should fulfill criteria for immediate provizionalization.
* Immediate insertion (e.g. placement of the implant immediately after extraction) will not constitute an exclusion criterion.
* The implants site(s) should be free from extraction remnants.
* The subject should be healthy and compliant with good oral hygiene.
* The subject should be available for the 5-year term of the investigation.
* Favorable and stable occlusal relationship

Exclusion Criteria:

* Alcohol or drug abuse as noted in patient records or in patient history.
* Health conditions, which do not permit the surgical procedure.
* Reason to believe that the treatment might have a negative effect on the subject's total situation (psychiatric problems), as noted in patient records or in patient history.
* The subject is not able to give her/his informed consent to participate.
* Any disorders in the planned implant area such as previous tumors, chronic bone disease, or previous irradiation.
* Severe bruxism or other destructive habits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2007-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Shorty Implants
Started | 38
Completed | 31
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Shorty Implants
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (4.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Marginal Bone Remodeling
Description: Marginal bone remodeling is calculated for each side of the implant (mesial and distal) separately, as the difference between bone levels at two time points. The average of mesial and distal remodeling is then calculated for each implant site (paired for each side between two different points). Negative numbers indicate bone loss. Implant insertion was defined as a baseline.
  Missing data was not imputed and not included in evaluation.
Time Frame: from implant insertion to 6, 12, 36 and 60 months
Population: Intention to treat analysis (all participants who received at least one implant were analyzed). Missing data was not imputed and not included in evaluation.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: implants
Groups:
- Shorty Implants: Brånemark System Mk III Shorty and NobelSpeedy Shorty
  Shorty implants: Dental implant insertion to maxilla or mandible
Arm/Group | Shorty Implants
Number analyzed (Participants) | 38
Number analyzed (implants) | 53
mm
  implant insertion to 6 months | -1.34 (1.10)
  implant insertion to 12 months | -1.38 (1.12)
  implant insertion to 36 months | -1.37 (1.02)
  implant insertion to 60 months | -1.65 (1.11)

2. Secondary Outcome: Cumulative Survival Rates of the Implants
Description: An implant was reported to be a surviving implant when it remained in the jaw and was functionally loaded even if not all the individual success criteria were fulfilled (i) an implant that causes no allergic, toxic or gross infectious reactions either locally or systemically, ii) offered anchorage to a functional prosthesis, iii) showed no signs of fracture or bending, iv) showed no signs of peri-implant radiolucency on an intraoral radiograph using a paralleling technique strictly perpendicular to the implant-bone interface, and v) showed no mobility when individually tested by either tapping or rocking with a hand instrument).
Time Frame: implant insertion to follow-up visits (6, 12, 36 and 60 months)
Population: as for outcome 1
Measure: Number; unit: percentage of surviving implants
Units Other Than Participants: implants
Arm/Group | Shorty Implants
Number analyzed (Participants) | 38
Number analyzed (implants) | 86
percentage of surviving implants
  60 months | 96.5
  36 months | 97.7
  12 months | 98.8
  6 months | 98.8

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the course of the study up to 5-years follow up.
Arm/Group | Shorty Implants
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 9/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Shorty Implants (N=38)
Implant mobile (Surgical and medical procedures) | 2 (2)
Implant Out (Surgical and medical procedures) | 2 (4)
Prosthesis retaining screw fracture (Surgical and medical procedures) | 1 (1)
Prosthesis retaining screw loosening (Surgical and medical procedures) | 3 (7)
Hyperplasia (Injury, poisoning and procedural complications) | 2 (2)
Swelling (Injury, poisoning and procedural complications) | 1 (1)
Moving quick temporary abutment (Surgical and medical procedures) | 1 (1)
Bridge loosening (Surgical and medical procedures) | 1 (1)
Phoenetic difficulties (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No